CLINICAL TRIAL: NCT05613725
Title: Optimising Laboratory Assays for Immune Responses to Gonococcus
Brief Title: OptiGon - Optimising Laboratory Assays for Immune Responses to Gonococcus
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OptiGon
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2022-11

CONDITIONS: Gonorrhea
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection

SUMMARY:
This is an observational study. Blood from otherwise healthy patients presenting with confirmed N.gonorrhoea infection, prior to treatment, will be collected to (i) allow the optimisation of assays assessing the immune response to gonococcus and (ii) assess whether N. gonorrhea specific responses can be detected on ELIspot +/- flow cytometry.

The investigators plan to recruit up to 30 adults (men and women, aged 18-50 years) who have been diagnosed with confirmed N.gonorrhoea infection at the Sexual Health Clinic at the Oxford University Hospitals NHS Foundation Trust. The investigators will collect blood samples from consenting participants prior to them receiving curative antibiotic treatment.

DETAILED DESCRIPTION:
On the day the patient attends the Sexual Health Clinic, they will be given the PIS to consider participation to the study following a confirmed positive result for N. gonorrhoea infection. Following written informed consent, a venous blood sample will be collected (up to 26 ml) on the same day. This will conclude that participant's involvement to the study.

The blood sample will be transported to the laboratory at the Jenner Institute, University of Oxford for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-50 years) attending Oxford University Hospitals NHS Foundation Trust with untreated confirmed N. gonorrhoea infection confirmed by either:

  * Nucleic acid test
  * Microscopy of urethral discharge

Exclusion Criteria:

* Have already received antimicrobial therapy to treat the N. gonorrhoea infection
* Have not provided written, informed consent.
* Presence of any known medical condition which, in the opinion of the local investigator, makes the donation of 26 mls of blood unsafe.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults (18-50 years) attending Oxford University Hospitals NHS Foundation Trust with confirmed untreated N. gonorrhoea infection
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Cellular immune response | Blood sampling at enrolment
  Cellular immune response detected by ELISpot +/- Flow cytometry from PBMCs collected from the blood of patients presenting with confirmed N.gonorrhoea infection.

CONTACTS AND LOCATIONS:
Overall Officials: Calman MacLennan, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom